CLINICAL TRIAL: NCT00200031
Title: Interstim Therapy Retrospective Cost Analysis and Quality of Life
Brief Title: A Cost Analysis of Interstim Therapy
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Other Study IDs: 4348
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Urinary Retention and Symptoms of Overactive Bladder (Urge, Frequency)
MeSH Terms: conditions — Urinary Retention

INTERVENTIONS:
Device: Interstim therapy

SUMMARY:
A study to examine the impact that Interstim Therapy for Urinary Control has on health care utilization and costs within a health care system and the satisfaction with treatment expressed by patients using this therapy.

DETAILED DESCRIPTION:
A retrospective administrative data analysis combined with a prospective health related quality of life/satisfaction with treatment survey designed to examine the impact that Interstim Therapy for Urinary Control has had on health care utilization and costs for the Kaiser Permanente system and the satisfaction with treatment expressed by patients using this therapy.

ELIGIBILITY:
Patients implanted with an Interstim Therapy for Urinary Control or undergoing test stimulation for potential placement of Interstim Therapy during the period of June 1, 2002 through June 30, 2004 and who are enrolled with Kaiser-Permanente of Southern California.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-07; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Aboseif, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Southern California Permanente Medical Group, Los Angeles, California, United States

REFERENCES:
- [Result] Aboseif SR, Kim DH, Rieder JM, Rhee EY, Menefee SA, Kaswick JR, Ree MH. Sacral neuromodulation: cost considerations and clinical benefits. Urology. 2007 Dec;70(6):1069-73; discussion 1073-4. doi: 10.1016/j.urology.2007.07.073. PMID 18158016